CLINICAL TRIAL: NCT03145792
Title: Online Coping Skills Counseling for Problem Gambling and Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Windsor (Other)
Collaborators: Manitoba Gambling Research Program (Unknown); Treatment Innovations (Industry); University of Manitoba (Other)
Responsible Party: Principal Investigator, David Ledgerwood, Adjunct Assistant Professor, University of Windsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-15-13
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Gambling Disorder; Trauma, Psychological; Problem Gambling; Posttraumatic Stress Disorder
MeSH Terms: conditions — Gambling; Psychological Trauma; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seeking Safety (Experimental): Behavioral therapy for trauma and addiction.
  Interventions: Behavioral: Seeking Safety
- CBT for Pathological Gambling (Active Comparator): Behavioral therapy for gambling problems.
  Interventions: Behavioral: CBT for Pathological Gambling

INTERVENTIONS:
Behavioral: Seeking Safety — Seeking Safety (SS) is a present-focused, evidence-based cognitive-behavioral therapy for trauma and/or addiction. It offers safe coping skills and education relevant to both problem areas.
  Arms: Seeking Safety
Behavioral: CBT for Pathological Gambling — Cognitive Behavior Therapy for Pathological Gambling (CBT-PG) is an evidence-based therapy for gambling problems. It focuses on cognitive correction, problem solving, social skills and relapse prevention.
  Arms: CBT for Pathological Gambling

SUMMARY:
This randomized controlled trial examines the efficacy of two behavioral therapies. Seeking Safety, which addresses co-occurring problem gambling (PG) and posttraumatic stress disorder (PTSD), is being compared to Cognitive-Behavioral Therapy for PG, which addresses only PG. Both models are delivered via telehealth.

DETAILED DESCRIPTION:
Our key study question is whether an integrated focus on PG and PTSD (Seeking Safety; SS) offers a useful new option for clinical care compared to a purely problem gambling approach (Cognitive-Behavioral Therapy for PG; CBT-PG). This question-the impact of integrated versus non-integrated treatment for co-occurring disorders-is one of the key issues in the field currently and has never been studied in relation to PG and PTSD.

Our aims are:

1. To conduct an RCT of SS versus CBT-PG in a sample of 84 people with current PG and PTSD (full or subthreshold).
2. To evaluate outcomes from baseline to end of treatment and 12 month followup on two primary variables (money lost gambling and number of gambling sessions) and several secondary variables.

Our hypotheses are: (a) SS will do no worse than CBT-PG on the primary PG outcomes as both treatments are designed to address addiction; i.e., both will show improvement from baseline to end of treatment and maintenance of gains through the followup. (b) SS will show superior results on trauma symptoms as SS is designed to address those, whereas CBT-PG is not.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Recruited from the province of Manitoba, Canada
* Meets criteria for PTSD (full or subthreshold) on the Clinician-Administered PTSD Scale (CAPS)
* Meets gambling disorder criteria per the DSM-5 Diagnostic Interview of Gambling Severity

Exclusion Criteria:

* Current uncontrolled psychotic or bipolar I disorder
* Suicidal or homicidal ideation with intent and/or plan
* Currently engaging in or planning to engage in any manualized, formal, evidence-based PTSD therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Money spent gambling | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Change from baseline in amount of money spent gambling in the past month
Number of gambling sessions | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Change from baseline in number of days in the past month during which gambling occurred

SECONDARY OUTCOMES:
PTSD Checklist (PCL) scores | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Posttraumatic stress disorder (PTSD) symptoms
Trauma Symptom Checklist 40 | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Change in baseline in broad trauma-related symptoms
Brief Symptom Inventory-18 scores | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Change from baseline in general psychiatric symptoms
Brief Addiction Monitor scores | 6-weeks (mid-treatment), 12-weeks (end-of-treatment), and 12-months
  Change from baseline in substance use and associated problems

CONTACTS AND LOCATIONS:
Overall Officials: David M Ledgerwood, PhD, Principal Investigator — University of Windsor; Lisa Najavits, PhD, Study Director — Treatment Innovations
Locations (1):
- Treatment Innovations, Newton Center, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided